CLINICAL TRIAL: NCT00378222
Title: A Prospective, Randomized Study of Single Versus Double Autologous Stem Cell Transplantation for Multiple Myeloma
Brief Title: Autologous Transplantation for Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO96
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Multiple Myeloma
Keywords: Myeloma previously untreated; Single autologous transplantation; Double autologous transplantation; Complete response
MeSH Terms: conditions — Multiple Myeloma; Pathologic Complete Response

INTERVENTIONS:
Procedure: Autologous Stem Cell Transplantation

SUMMARY:
The present study was designed in an attempt to prospectively evaluate in a randomized fashion whether further cytotoxic dose intensification, as delivered with two sequential autologous stem-cell transplantations, improved the outcome of younger patients with newly diagnosed multiple myeloma in comparison with a single autologous transplantation.

DETAILED DESCRIPTION:
Following demonstration that single autologous transplantation for the treatment of younger patients with newly diagnosed multiple myeloma prolonged overall survival in comparison with conventional chemotherapy, double autologous transplantation was tested, initially in refractory myeloma and subsequently to include also patients with newly diagnosed disease. To explore the role of double autologous stem-cell transplantation as part of up-front therapy for multiple myeloma, in 1996 we launched a prospective, randomized trial comparing a single course of stem-cell-supported melphalan with the same regimen followed, after three to six months, by a second autologous transplantation in support of melphalan and busulfan. The study was designed to detect a 15 percent increase in complete or near complete response rate with double transplants compared to a single transplantation. With a 2-sided significance level α = 0.05 and a power 1-β = 0.80, 162 patients were required in each treatment arm of the study to detect a statistically significant increase in complete or near complete response rate from 30% in the single-transplant arm to 45% in the double-transplant arm. Primary study endpoint was the complete or near complete response rate. Secondary study endpoints were relapse-free survival, event-free survival and overall survival. The recruitment target was 324 patients.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated
* Younger than 61 years
* Symptomatic myeloma
* Measurable disease
* Fit to receive high-dose chemotherapy

Exclusion Criteria:

* M-GUS
* Solitary plasmacytoma
* Plasma cell leukemia
* AL Amyloidosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 324
Dates: Start 1996-01; Study Completion 2005-11

PRIMARY OUTCOMES:
Complete or near Complete Response Rate

SECONDARY OUTCOMES:
Relapse-free Survival
Event-free Survival
Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Michele Cavo, MD, Principal Investigator — Institute of Hematology and Medical Oncology - University of Bologna

REFERENCES:
- [Result] Cavo M et al. Superiority of Double over Single Autologous Stem Cell Transplantation as First-Line Therapy for Multiple Myeloma. Blood (ASH Annual Meeting Abstracts) 2004 104: Abstract 536